CLINICAL TRIAL: NCT03335319
Title: The Effect Of An Expanded Long Term Periodization Exercise Training In Patients With Cardiovascular Disease: Central And Peripheral Adaptations
Brief Title: The Effect Of An Expanded Long Term Periodization Exercise Training In Patients With Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Maria Helena Santa-Clara Pombo Rodrigues, Assistant Professor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 30/2017
Record Dates: First submitted 2017-10-22; First posted 2017-11-07 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Cardiovascular Disease; Coronary Artery Disease; Cardiopulmonary Exercise Testing; Oxygen Uptake Kinetics; Skeletal Muscle Oxygenation; Exercise Training; Periodized Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomized and stratified (by gender and age) into either one of the two groups exercise training groups: 1) periodization or 2) non periodization. The randomization code will be developed with a computer random-number generator to select random permuted blocks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodized Exercise Training Regime (Experimental): The ET program will be carried out 3 times a week (60 minutes per session) on non-consecutive days for 48 weeks and supervised for both groups. Exercise prescription will be gradually progressed through various combinations of duration, frequency and/or intensity of training. Over the 1st-15th exercise sessions: MCT and anatomical resistance training; from the 16th-30th session: combined ET with HIIT and hypertrophy; from the 31st-45th exercise session, after the adjustments of the respectively time point assessments: MCT and maximal strength; from the 46th-60th exercise sessions: HIIT with hypertrophy; at the end of the 60th session until the end (6 months has passed): the same exercise prescription will repeat all over again at the same order.
  Interventions: Other: Periodized Exercise Training Regime
- Non Periodized Exercise Training Regime (Active Comparator): participants will do a combined ET regime (aerobic and RT). Aerobic component: combine moderate to vigorous exercises 3 d.wk-1 on nonconsecutive days, for 20 min per session, involving major muscle groups using the available ergometers to perform continuous and rhythmic activities in nature. Resistance component: RT should be performed after the aerobic component of the exercise session to allow for adequate warm-up. Initial load should be trained initially with one set of 10-15 repetitions that can be lifted without straining (~30%-40% 1RM for the upper body; ~50%-60% 1 RM for the lower body). Each major muscle group should be trained initially with one set; multiple set regimens may be introduced later as tolerated. It will be performed 8-10 exercises of the major muscle groups.
  Interventions: Other: Non Periodized Exercise Training Regime

INTERVENTIONS:
Other: Periodized Exercise Training Regime — MCT 1st: 20 min on an ergometer; at Anaerobic Threshold (AT) 1 or, if the AT could not be adequately determined, 50-60% of the Heart Rate Reserve (HRR), Borg Rating of Perceived Exertion (RPE) equivalent 9-11. MCT 2nd: 20 minutes; 60-70%HRR, RPE 12-13. HIIT 1st: 4 interval training periods of 2 minutes (AT2 intensity or 80-90%HRR, RPE 15-17) and 4 active pauses of 2 minutes (below AT 1 or 40-50%HRR, RPE 6-9) between interval training periods. HIIT 2nd: same intervals as in 1st HIIT different intensities: high intensity interval above AT2 intensity or > 90%HRR, RPE 17-19 and active pauses at AT 1 or 50-60%HRR, RPE 9-11. Resistance training adaptation: 2 sets of 15-20 repetitions 50% 1RM; Hypertrophy: 2 sets 8-12 repetitions at 60% 1RM; Maximal Strength: 2 sets of 6-8 repetitions at 80% 1RM.
  Arms: Periodized Exercise Training Regime
Other: Non Periodized Exercise Training Regime — To ensure that total training loads were similar in both groups despite differences in intensity, it will be used the training impulses (TRIMP) method from Edwards for the aerobic component and the volume load method for the RT component. All sessions will include 10 minutes of warm up and cool down standardized for both groups. By design, the non periodized group involves an identical total training volume and time commitment but differed regarding metabolic stress induced by the linear periodized group. All patients will be monitored with a HR monitor during the execution of the exercise session in order to achieve the HR training. Blood pressure will be assessed before and after completing each session. If necessary, the blood pressure will be measured during the ET session.
  Arms: Non Periodized Exercise Training Regime

SUMMARY:
Benefits from cardiac rehabilitation (CR) programs are evidence based and widely recognized. Less than 50% of people who participate in hospital-based CR programs maintain an exercise regimen for as long as six months after completion. Despite the benefits associated with regular exercise training (ET), adherence with supervised exercise-based CR remains low.

Current exercise guidelines for CR focus on moderate intensity steady state exercises, with walking and cycling being the most recommended types of ET. The repetitive nature of this type of activity can become monotonous for the patient, affecting exercise adherence, compliance and training outcomes. Exercise periodization is a method typically used in sports training, but the impact of periodized exercise to yield optimal beneficial effects in cardiac patients is still unclear.

In healthy or trained populations, periodization aims to optimize ET adaptations as compared with non periodized training, to prevent overtraining and to avoid plateauing of training adaptations. Periodized methods are considered to be superior to non periodized methods in trained populations and appears to be superior in inactive adults. In most of the CR programs there are no periodization or exercise progression during medium to long term interventions. Further randomized controlled trials (RCT) are necessary to evaluate long-term periodization outcomes.

The purpose of this research project is twofold:

1. To conduct a 12-month randomized control trial to evaluate the effects of a periodized ET regime versus a non periodized ET regime (guidelines) on VO2 peak, maximal strength, body composition, functionality and quality of life in cardiovascular disease patients.
2. to differentiate the effects of a 12-month periodized ET regime versus a non periodized ET regime on the different components of the oxygen kinetics response and oxidative adaptations in cardiovascular disease patients.

These patients will be randomized in 2 ET groups: 1) periodization; 2) non periodization. This experimental design will occur during 48 weeks 3 times per week with 4 assessment time points: M0) before starting the ET program (baseline); M1) 3 months after starting the ET; M2) 6 months after starting the ET program and M3) 12 months at the end of the community-based ET program.

DETAILED DESCRIPTION:
Cardiac Rehabilitation (CR) of patients with Cardiovascular Disease (CVD) has been practiced in Europe to varying degrees since the early 1970s. CR is a comprehensive, long-term program involving medical evaluation, prescribed Exercise Training (ET), cardiac risk factor modification, education and counselling. These programs are designed to limit the physiologic and psychological effects of cardiac illness, reduce the risk for sudden death or re-infarction, control cardiac symptoms, stabilize or reverse the atherosclerotic process, and enhance the psychosocial and vocational status of selected patients. Furthermore, it is a safe, useful and an effective treatment for patients with coronary artery disease (CAD), particularly after myocardial infarction, but also for patients with cardiac interventions and chronic stable heart failure.

Exercise adherence after a hospital-based CR program is reported to be poor with only 30% to 60% of those who complete a phase II CR program are still exercising 6 months later and after 12 months, up to 50 to 80% of participants failing to adhere to exercise. Despite the benefits associated with regular ET, adherence with supervised exercise-based CR remains low.

A brief review of meta-analysis studies that assess the impact of different types of exercise in short term outcomes for participants of CR will now be presented. The findings of a meta-analysis in 2015 indicated that high intensity interval training (HIIT) is more effective than moderate continuous training (MCT) for the improvement of both VO2 peak and the anaerobic threshold in patients with stable CAD. The greater improvement in VO2 peak following HIIT compared to MCT (4.6 ± 3.1 versus 2.8 ± 2.4 ml/kg/min) is important in the context of a 10-25% survival advantage with every 3.5 ml/kg/min improvement in VO2 peak.

Another meta-analysis in 2016, compared HIIT and MCT in their ability to improve patients aerobic exercise capacity and various cardiovascular risk factors. Ten studies with 472 patients were included for analyses (218 HIIT, 254 MCT) and the main conclusions were that HIIT improves the mean VO2 peak in patients with CAD more than MCT, although MCT was associated with a more pronounced numerical decline in patients resting heart rate and body weight.

Current CR guidelines recommend the inclusion of a standardized resistance training (RT) program. A recent meta-analysis of ET programs in patients with CAD revealed that the addition of RT training to MCT led to superior improvements in body composition, muscle strength, peak work capacity, and a trend for greater increases in VO2 peak. Similar to HIIT, RT has not been shown to compromise patient safety or program adherence.

Less is known about central and peripheral adaptations during long term effects on HIIT, MCT or even aerobic combined training with RT. In 2016, a systematic review and meta-analysis with a total of 63 studies with 14,486 participants with CAD median follow-up of 12 months were included. It was concluded that exercise-based CR reduces cardiovascular mortality and provides important data showing reductions in hospital admissions and improvements in quality of life. Madssen et al, showed that a 12-month maintenance exercise program consisting of infrequent supervised exercise sessions did not result in improved adherence to exercise or increased VO2 peak in CAD patients compared to usual care. One monthly session during a year of HIIT was not enough to improve or maintain exercise capacity. In the literature there is a lack of evidence on the effects in exercise capacity, muscle strength and body composition in long term weekly supervised exercise sessions on a maintenance exercise program in CVD patients.

Current exercise guidelines for CR focus on moderate intensity steady state exercises, with walking and cycling being the most recommended types of ET. Multiple training variables can be manipulated during exercise prescription, including repetitions, interval length, rest period length and intensity of resistance. In this regard, much insight could be gained from approaches used in sport conditioning, where exercise prescription is designed to be physiologically and psychologically sustainable using periodization.

Periodization is defined as an organized cyclic program that uses planned variations in intensity, volume, and specificity to minimize fatigue and maximize performance outcomes. In healthy or trained populations, periodization aims to optimize ET adaptations as compared with non periodized training, to prevent overtraining and to avoid plateauing of training adaptations. Periodized methods are considered to be superior to non periodized methods in trained populations and appears to be superior in inactive adults. Interestingly, a recent study investigated the effect of 22 weeks of 2 different types of periodization and non periodization resistance training protocols on a comprehensive range of physical function and health outcomes in apparently healthy untrained older adults. Contrary of what was hypothesised, all three training models were equally effective for promoting significant improvements in various physical function and physiological health outcomes through resistance training in this population.

In most of the CR programs there are no periodization or exercise progression during medium to long term interventions. Evaluate long-term periodization outcomes and assess the length of change observed in supervised CR programs might be of interest and necessary.

This study will hopefully contribute to generate evidence-based exercise prescription approaches to prolong the ET after the end of hospital-based CR programs.

The purpose of this research project is twofold:

1. To conduct a 12-month randomized control trial to evaluate the effects of a periodized ET regime versus a non periodized ET regime (guidelines) on VO2 peak, maximal strength, body composition, functionality and quality of life in CVD.
2. to differentiate the effects of a 12-month periodized ET regime versus a non periodized ET regime on the different components of the oxygen kinetics response and oxidative adaptations in CVD patients.

The hypothesis for this study are: 1) considering that this type of periodization exerts higher stress on the cardiovascular and neuromuscular systems, so that there could be greater adaptations leading to higher increases in VO2max, muscle strength, body composition and functionality compared to non periodized ET regime; 2) there will be a better improvement microvascular O2 delivery in the exercise transient in response to periodized ET regime that will be associated with a faster adjustment of pulmonary VO2 kinetics than in non periodized group. Improvements in microvascular O2 delivery will be indicated by a better matching between the rate of adjustment of muscle deoxygenation relative to phase II pulmonary VO2, which represents a decreased reliance on O2 extraction for a given pulmonary VO2.

STUDY DESIGN:

A longitudinal RCT research design performed in the Cardiovascular Rehabilitation Center of the University of Lisbon (CRECUL) at the Lisbon University Stadium (EUL) using two distinct ET prescriptions (periodization vs non periodization) will be applied in cardiovascular disease patients. Briefly, following the informed consent process, patients will be randomized and stratified (by gender and age) to periodization or non periodization groups. The randomization code will be developed with a computer random-number generator to select random permuted blocks. Participants will exercise for a period of 12 months. All the same assessments, except the echocardiogram that will be done in M0 and M3 (for risk stratification), are going to be taken in 4 different time points during a year: M0 - baseline, M1 - 3 months after starting the ET, M2 - 6 months after starting the ET and M3 - 12 months after starting the ET. The patients will be randomized into either one of the two ET group.

Sample size was calculated (G-Power, Version 3.1.3) assuming a difference in peak oxygen uptake (VO2 peak) between groups of 3 ml/kg/min to be a clinical important difference with a standard deviation of 3.5 ml/kg/min, α=0.05, 1-β=0.80 and an expected dropout rate of 50%. The calculations yielded a total minimum sample size of 56 participants (28 in each group).

The following assessments on the 4 time points will be performed at the Pulido Valente Hospital, Faculty of Human Kinetics - University of Lisbon (FMH-UL) and Academia de Fitness at EUL: Echocardiogram (Echo) (MyLab Alpha, ESAOTE); cardiopulmonary exercise test (CPET) (Ergostik, Geratherm Respiratory GmbH, Bad Kissingen); skeletal muscle deoxygenation dynamics (NIMO, Nirox srl); body composition - dual energy radiographic absorptiometry (DXA, Hologic Explorer-W); objective measured physical activity - accelerometer (ActiGraph GT3X+); functional physical fitness - Fullerton Functional Fitness Test; isometric strength - portable hand dynamometer JAMAR plus digital (Sammons Preston); maximal strength - 1RM and Quality of Life questionnaire (Short Form-36 Health Survey).

All assessment moments will be done in 1 to 2 weeks:

Day 1 - Echo and CPET will be performed at the Hospital; Day 2 and 3 - during the day and time of the ET session at the EUL, the patient will perform: functional physical fitness tests; maximal strength; isometric strength and Quality of Life questionnaire; Day 4 - In FMH-UL, the dual energy radiographic absorptiometry (DXA) exam and the activation of the accelerometer to measure the objective measured physical activity will be done.

Day 5 - Submaximal CPET with the skeletal muscle deoxygenation dynamics at the Hospital.

In order to assure the confidentiality of the participants an ID code will be attributed to each participant in the database and all the equipment's and sheets used. A single researcher will perform the database management.

DATA ANALYSIS:

Data will be analyzed in M0, M1, M2 and M3. It will be tested the data for normality and homogeneity of variance with the Shapiro Wilk and Levene's tests, respectively. Data analysis will be described according to the established purposes for this project (descriptive values: mean, standard deviation, range, % change) and comparisons of means will be used for all purposed outcomes intra and inter groups. Baseline characteristics between groups will be evaluated with oneway ANOVA. Mixed between within subjects ANOVA will be conducted in a 2 (pre vs post ET) design to assess efficiency of the program. When a significant interaction is observed, t tests, or Wilcoxon signed-rank tests will be used to determine where the interaction occurred.

M0 versus M1, M0 versus M2, M0 versus M3, M1 versus M2, M2 versus M3 and M1 versus M3 will be compared to evaluate the changes in patients and trace the necessary timespan for such changes using General Linear Mixed Model Analysis for repeated measures with Tukey's post hoc procedure for the mean comparisons. Pearson product moment correlation coefficient or Spearman's rank correlation coefficient will be used to study the relationship between different variables by group and correlation coefficients will be compared between groups. Statistical significance will be set at an alpha level of 0.05. Other statistical procedures can be done.

Statistical analyses will be conducted using Statistical Package for the Social Sciences (SPSS) 22.0 (IBM SPSS Statistics, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* angiographically documented coronary artery disease in at least one major epicardial vessel
* myocardial infarction,
* coronary revascularization (coronary artery bypass grafting, percutaneous transluminal coronary angioplasty, or coronary artery stent),

Exclusion Criteria:

* heart failure
* unstable angina pectoris
* heart transplants with either cardiac resynchronization therapy or implantable defibrillators
* inability to comply with guidelines for participation in exercise testing and training
* significant limiting and/or unstable comorbidities that would prevent full participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change of peak oxygen consumption during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  A symptom-limited ramp incremental cardiopulmonary exercise test, will be performed on a cycle ergometer (Ergostik, Geratherm Respiratory GmbH, Germany) with breath-by-breath gas exchange measurements. Each patient will be encouraged to exercise to exhaustion (20 Watt+20 Watt/min or 15 Watt+15 Watt/min or 10 Watt+10 Watt/min), as defined by intolerance, leg fatigue or dyspnea unless clinical criteria for test termination occurred. Peak oxygen capacity will be considered the highest attained VO2 during the final 30s of exercise. All patients should achieve a respiratory exchange ratio of >1.1, an indicator of maximal effort.
Change of oxygen kinetics during submaximal test | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The test load is set at 80% of the value of the work rate corresponding to the Anaerobic Threshold detected in the maximum test, which was performed first, or 50% of VO2 peak, if the Anaerobic Threshold could not be adequately determined. Cardiopulmonary data will be recorded for 5 minutes at rest followed by 1 minute unloaded pedaling. After unloaded pedaling, patients will perform the constant load test for 6 min at the work rate described above, followed by unloaded pedaling for 5min. To improve the confidence of the kinetic parameter determination, this test will be performed three times and the averaged profile will be used for the kinetic analysis.

SECONDARY OUTCOMES:
Change of Anaerobic Threshold VO2 during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Change in VO2 reached at the maximal cardiopulmonary exercise test at the Anaerobic Threshold.
Change of Anaerobic Threshold Heart Rate during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Change in heart rate reached at the maximal cardiopulmonary exercise test at the Anaerobic Threshold.
Change of Anaerobic Threshold Watts during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Change in watts reached at the maximal cardiopulmonary exercise test at the Anaerobic Threshold.
Change of Respiratory Compensation Point VO2 during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Change in VO2 reached at the maximal cardiopulmonary exercise test at the Respiratory Compensation Point.
Change of Respiratory Compensation Point Heart Rate during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Change in heart rate reached at the maximal cardiopulmonary exercise test at the Respiratory Compensation Point.
Change of Respiratory Compensation Point Watts during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Change in watts reached at the maximal cardiopulmonary exercise test at the Respiratory Compensation Point.
Change of Peak Heart Rate reached during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Maximal heart rate reached at the cardiopulmonary exercise testing.
Change of Maximal Watts reached during cardiopulmonary exercise testing | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Maximal watts reached at the cardiopulmonary exercise testing.
Change of Deoxyhaemoglobin of the vastus lateralis muscle at the submaximal test | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The muscle deoxygenation dynamics of the Vastus Lateralis muscle will be evaluated throughout the submaximal CPET. Deoxyhaemoglobin (HHb) concentration will be quantified with a continuous-wave tissue oximeter (NIMO, Nirox srl, Brescia, Italy), based on the Near-infrared Spectroscopy (NIRS) system, which provides continuous, non-invasive monitoring of the relative concentration changes in these variables during rest and exercise.
Change of Oxyhaemoglobin of the vastus lateralis muscle at the submaximal test | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The muscle deoxygenation dynamics of the Vastus Lateralis muscle will be evaluated throughout the submaximal CPET. Oxyhaemoglobin (HbO2) concentration will be quantified with a continuous-wave tissue oximeter (NIMO, Nirox srl, Brescia, Italy), based on the Near-infrared Spectroscopy (NIRS) system, which provides continuous, non-invasive monitoring of the relative concentration changes in these variables during rest and exercise.
Change of Total Haemoglobin of the vastus lateralis muscle at the submaximal test | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The muscle deoxygenation dynamics of the Vastus Lateralis muscle will be evaluated throughout the submaximal CPET. Total haemoglobin (HbT) concentration will be quantified with a continuous-wave tissue oximeter (NIMO, Nirox srl, Brescia, Italy), based on the Near-infrared Spectroscopy (NIRS) system, which provides continuous, non-invasive monitoring of the relative concentration changes in these variables during rest and exercise.
Change of Maximal Strength | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Maximal strength will be assessed by 1 Repetition Maximum (1RM) test for each of six weight exercises on variable resistance machines as follows: leg press, leg extension, leg curl, low row, chest press and lat pull down. The protocol will include four pre-test sessions to familiarize each patient with the test procedures. Correct exercise and breathing techniques (avoidance of the Valsalva manoeuvre) will be practiced.
Change of Lean Soft-Tissue | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Total and regional lean soft-tissue will be estimated using dual energy radiographic absorptiometry (DXA) (Hologic Explorer-W, fan-beam densitometer, software QDR for windows version 12.4, Hologic, USA).
Change of Fat Mass | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Total and regional body mass fat mass will be estimated using dual energy radiographic absorptiometry (DXA) (Hologic Explorer-W, fan-beam densitometer, software QDR for windows version 12.4, Hologic, USA).
Change of Bone Mineral Content | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  Total bone mineral content will be estimated using dual energy radiographic absorptiometry (DXA) (Hologic Explorer-W, fan-beam densitometer, software QDR for windows version 12.4, Hologic, USA).
Change of Quality of Life | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The Short Form-36 Health Survey (SF-36) is a self-assessment health status questionnaire composed of 36 questions about socio-demographic, health and personal behavior. A Portuguese validated version of SF-36 is available.

OTHER OUTCOMES:
Change of six minute walking test distance | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The six minute walking test (6MWT) will be performed indoors, along a long flat, straight, enclosed 20-meter corridor with a hard surface that is seldom. Total distance during the test will be recorded.
Change of 30-second chair stand repetitions | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The 30-second chair stand, assesses the lower body strength, needed for numerous tasks such as climbing stairs or walking.
Change of 8-foot up and go test duration | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  The 8-foot (2.44 meters) up and go test evaluates the agility/dynamic balance, which is important in tasks that require quick maneuvering.
Change of chair sit-and-reach distance reached | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  For the flexibility for the lower limbs it will be assessed the chair sit-and-reach.
Change of back scratch test distance reached | At baseline, 3 months after starting the ET, 6 months after starting the ET and 12 months after starting the ET
  For the flexibility for the upper limbs it will be assessed the back scratch test.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Santa-Clara, PhD, Principal Investigator — Faculty of Human Kinetics, University of Lisbon
Locations (1):
- Faculty of Human Kinetics - University of Lisbon, Lisbon, Cruz Quebrada, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Participant data for all primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Humphrey R, Guazzi M, Niebauer J. Cardiac rehabilitation in Europe. Prog Cardiovasc Dis. 2014 Mar-Apr;56(5):551-6. doi: 10.1016/j.pcad.2013.08.004. Epub 2013 Oct 5. PMID 24607021
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Elliott AD, Rajopadhyaya K, Bentley DJ, Beltrame JF, Aromataris EC. Interval training versus continuous exercise in patients with coronary artery disease: a meta-analysis. Heart Lung Circ. 2015 Feb;24(2):149-57. doi: 10.1016/j.hlc.2014.09.001. Epub 2014 Sep 16. PMID 25306500
- [Background] Liou K, Ho S, Fildes J, Ooi SY. High Intensity Interval versus Moderate Intensity Continuous Training in Patients with Coronary Artery Disease: A Meta-analysis of Physiological and Clinical Parameters. Heart Lung Circ. 2016 Feb;25(2):166-74. doi: 10.1016/j.hlc.2015.06.828. Epub 2015 Jul 22. PMID 26375499
- [Background] Marzolini S, Oh PI, Brooks D. Effect of combined aerobic and resistance training versus aerobic training alone in individuals with coronary artery disease: a meta-analysis. Eur J Prev Cardiol. 2012 Feb;19(1):81-94. doi: 10.1177/1741826710393197. Epub 2011 Feb 21. PMID 21450617
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Madssen E, Arbo I, Granoien I, Walderhaug L, Moholdt T. Peak oxygen uptake after cardiac rehabilitation: a randomized controlled trial of a 12-month maintenance program versus usual care. PLoS One. 2014 Sep 23;9(9):e107924. doi: 10.1371/journal.pone.0107924. eCollection 2014. PMID 25247991
- [Background] Rhea MR, Alderman BL. A meta-analysis of periodized versus nonperiodized strength and power training programs. Res Q Exerc Sport. 2004 Dec;75(4):413-22. doi: 10.1080/02701367.2004.10609174. PMID 15673040
- [Background] Strohacker K, Fazzino D, Breslin WL, Xu X. The use of periodization in exercise prescriptions for inactive adults: A systematic review. Prev Med Rep. 2015 May 6;2:385-96. doi: 10.1016/j.pmedr.2015.04.023. eCollection 2015. PMID 26844095
- [Background] Conlon JA, Newton RU, Tufano JJ, Banyard HG, Hopper AJ, Ridge AJ, Haff GG. Periodization Strategies in Older Adults: Impact on Physical Function and Health. Med Sci Sports Exerc. 2016 Dec;48(12):2426-2436. doi: 10.1249/MSS.0000000000001053. PMID 27434088
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Yamamoto S, Hotta K, Ota E, Mori R, Matsunaga A. Effects of resistance training on muscle strength, exercise capacity, and mobility in middle-aged and elderly patients with coronary artery disease: A meta-analysis. J Cardiol. 2016 Aug;68(2):125-34. doi: 10.1016/j.jjcc.2015.09.005. Epub 2015 Dec 12. PMID 26690738
- [Background] Shepherd CW, While AE. Cardiac rehabilitation and quality of life: a systematic review. Int J Nurs Stud. 2012 Jun;49(6):755-71. doi: 10.1016/j.ijnurstu.2011.11.019. Epub 2011 Dec 23. PMID 22197653
- [Derived] Pinto R, Angarten V, Santos V, Melo X, Santa-Clara H. The effect of an expanded long-term periodization exercise training on physical fitness in patients with coronary artery disease: study protocol for a randomized controlled trial. Trials. 2019 Apr 11;20(1):208. doi: 10.1186/s13063-019-3292-9. PMID 30975195
- See also: Official Website of the Cardiovascular Rehabilitation Center of the University of Lisbon (CRECUL) — https://www.estadio.ulisboa.pt/info/centro-de-reabilitacao-cardiovascular

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT03335319/Prot_SAP_001.pdf